CLINICAL TRIAL: NCT01807624
Title: The Pharmacokinetics Of Tetracaine, Para-Butylaminobenzoic Acid, And Oxymetazoline After Intranasal Administration Of The Highest Phase 3 Dose Of Kovacaine™ Mist To Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of Kovacaine Nasal Spray (24 Hour Blood Collection)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Triligent International (Industry); Rho, Inc. (Industry); Analytical Bio-Chemistry Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR 2-06
Record Dates: First submitted 2013-03-05; First posted 2013-03-08 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
Keywords: Pharmacokinetic
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kovacaine Mist (Experimental): Tetracaine HCl 3% and Oxymetazoline HCl 0.05% - 3 sprays will be administered at the start of the procedure
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%

INTERVENTIONS:
Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% — 1 spray is 0.2mL is volume and contains 6mg Tetracaine HCl 3% and 0.1mg Oxymetazoline HCl (para-butylaminobenzoic acid or PABA is active metabolite)
  Other Names: Kovacaine Nasal Spray

SUMMARY:
The purpose of this study is to determine the pharmacokinetics/pharmacodynamics and safety of a nasal spray containing the anesthetic drug tetracaine in combination with oxymetazoline with blood draws over 24 hours.

DETAILED DESCRIPTION:
The purpose of this study is to determine the pharmacokinetics and safety of tetracaine, para- butylaminobenzoic acid (PBBA), and oxymetazoline after intranasal administration of the highest Phase 3 dose of Kovacaine Mist (Tetracaine Hydrochloride with Oxymetazoline Hydrochloride) to healthy volunteers.

This is an open-label, single-treatment, single-dose study in healthy volunteers in which all subjects will receive the highest Phase 3 dose of Kovacaine Mist on one occasion. No randomization is necessary for this single treatment, single dose study. A single study center will participate.

Each subject will receive a single dose of Kovacaine Mist (3% tetracaine HCl with 0.05% oxymetazoline HCl) consisting of 3 sprays (each 0.2 mL) in one nostril not taking longer than 8 minutes, for a total 0.6 mL dose containing 18 mg tetracaine HCl and 0.3 mg oxymetazoline HCl.

The total dosing period will be 8 minutes. Subjects will be required to fast 10 hours prior to dosing and for four (4) hours after dosing. Water will be allowed ad lib during the study except for one (1) hour prior through one (1) hour after dose administration. Subjects will be admitted to the study unit no later than 2100 hours of the evening prior to drug administration and will remain in the unit until the 24 hour blood sample is collected and discharge procedures are completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breast-feeding female subjects between the ages of 18 and 75 years (inclusive).
* Can understand and sign the informed consent document, can communicate with the investigator, and can understand and comply with the requirements of the protocol.
* Body mass index between 18 and 35 BMI.
* Sufficiently healthy as determined by the investigator to receive the test medications and undergo the scheduled study procedure.
* Can breathe through both nostrils.
* Screening BP ≤ 140/90 mm Hg.

Exclusion Criteria:

* History of clinically significant respiratory, gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, including cardiac arrhythmia, narrow angle glaucoma and benign prostatic hypertrophy (in men), uncontrolled thyroid disease (including Hashimoto's Thyroiditis and lymphocytic thyroiditis), uncontrolled diabetes mellitus or any other condition which, in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Has clinically significant abnormal findings on the physical examination, medical history, electrocardiogram (ECG), or clinical laboratory evaluation during screening. This includes current upper respiratory infections.
* Currently experiencing seasonal or perennial allergic rhinitis, recurrent nose-bleeds or asthma, or has a significant history of these conditions, in the opinion of the Investigator.
* Current, including the last 30 days, sinusitis or other upper respiratory infections.
* Nasal polyps, significant nasal or sinus surgery or other abnormality that may interfere with the dose administration.
* History of allergic or adverse responses to tetracaine, other ester local anesthetics, PBBA, oxymetazoline and its preservatives, or para-aminobenzoic acid as found in PABA containing sunscreens or any comparable or similar product.
* Donation of blood or plasma within 30 days of the first dose of Study Drug.
* Participation in a clinical trial within 30 days prior to the first dose of Study Drug.
* Use of any new over-the-counter (OTC) medication, including topical anesthetic creams or gels, vitamins, within seven days prior to the first dose of the Study Drug or during the study unless approved by the Principal Investigator.
* Any prescription medication, whose dose is not stable at the time of screening, as determined by the Principal Investigator.
* Treatment with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of Study Drug or during the study.
* Smoking or use of tobacco products within 6 months prior to the first dose of Study Drug or during the study.
* Female trying to conceive, is pregnant, suspected of being pregnant, or is lactating. (Females of child-bearing potential will be required to take a serum pregnancy test at screening (up to 21 days prior to the start of the study, including the day of the study), as well as a urine pregnancy test at check-in to rule out pregnancy.)
* Positive serum pregnancy test at screening or urine pregnancy test at check-in for all women of childbearing potential.
* Positive blood screen for HIV, Hepatitis B surface antigen (HbSAg), or Hepatitis C, or a positive urine screen for alcohol, drugs of abuse, or cotinine.
* Have a history of pseudocholinesterase deficiency or previous prolonged paralysis with succinylcholine or difficulty waking up from general anesthesia.
* Have a history of alcoholism and/or drug abuse.
* Have taken a monoamine oxidase inhibitor or vasopressor drug within the past 3 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Mulvahill, Study Chair — St. Renatus
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Kovacaine Nasal Spray: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% - 3 sprays will be administered at the start of the procedure
  Tetracaine HCl 3% and Oxymetazoline HCl 0.05%: 1 spray is 0.2mL is volume and contains 6mg Tetracaine HCl 3% and 0.1mg Oxymetazoline HCl
Period: Overall Study
Arm/Group | Kovacaine Nasal Spray
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 19
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Oxymetazoline and PBBA
Time Frame: 0, 5, 10, 15, 20, 25, 30, 40, 50 minutes, and 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours after completion of the last nasal spray
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
ng/mL
  Oxymetazoline | 1.79 (0.586)
  PBBA | 465 (122)

2. Primary Outcome: Tmax of Oxymetazoline and PBBA
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
minutes
  Oxymetazoline | 5.8 (1.9)
  PBBA | 22 (6.6)

3. Primary Outcome: Half-life of Oxymetazoline and PBBA
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
minutes
  Oxymetazoline | 5.23 (2.2)
  PBBA | 2.6 (1.23)

4. Primary Outcome: AUC0-t of Oxymetazoline and PBBA
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
ng*h/mL
  Oxymetazoline | 3.67 (1.79)
  PBBA | 960 (509)

5. Primary Outcome: AUC0-infinity of Oxymetazoline and PBBA
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
ng*h/mL
  Oxymetazoline | 4.24 (2.09)
  PBBA | 973 (513)

6. Secondary Outcome: Increase in SBP > 20 mmHg on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 3

7. Secondary Outcome: Decrease in SBP > 20 mmHg on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 0

8. Secondary Outcome: Increase in DBP > 20 mmHg on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 1

9. Secondary Outcome: Decrease in DBP > 20 mmHg on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 0

10. Secondary Outcome: Increase in Pulse Rate > 20 Bpm on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 2

11. Secondary Outcome: Decrease in Pulse Rate > 20 Bpm on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 2

12. Secondary Outcome: SpO2 Increase of > 5% on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 0

13. Secondary Outcome: SpO2 Decrease of > 5% on 2 Consecutive Measurements After Administration of Study Medication
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 24
participants | 0

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Kovacaine Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 22/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Nasal Spray (N=24)
Nausea (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 11 — Runny nose
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No